CLINICAL TRIAL: NCT02531230
Title: "All Comers" Post Market Clinical Follow-up (PMCF) With Multi-LOC for flOw liMiting Outcomes After Plain Old Balloon Angioplasty (POBA) and/or Drug Coated Balloon (DCB) Treatment in the Infra-inguinal Position With the objectiVE to Implant Multiple Stent Segments
Brief Title: "All Comers" Post Market Clinical Follow-up (PMCF) With Multi-LOC for flOw liMiting Outcomes
Acronym: LOCOMOTIVE
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: Deaconess Hospital Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1502
Record Dates: First submitted 2015-05-29; First posted 2015-08-24 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VascuFlex Multi-LOC® — Multi-LOC® peripheral stent system for bailout stenting after Plain Old Balloon Angioplasty (POBA) or Drug Coated Balloon (DCB) Angioplasty

SUMMARY:
The aim of the study is to assess the safety and efficacy of the Multi-LOC® peripheral stent system to treat de novo and restenotic lesions (no in-stent restenosis (ISR), no restenosis post drug coated balloon (DCB) after flow limiting plain old balloon angioplasty (POBA) and/or DCB dilatations in the superficial femoral artery (SFA) and popliteal segments (P1, P2 & P3)

DETAILED DESCRIPTION:
This study is an non-randomized, prospective, multi-center, non-interventional study (registry, for Germany: §23b MPG)

ELIGIBILITY:
Inclusion Criteria:

* Willingness to treat flow-limiting dissections/recoil after plain old balloon angioplasty (POBA)/drug coated balloon (DCB) interventions
* Patients in Rutherford classes 2 through 5
* Patients eligible for peripheral revascularization by means of percutaneous transluminal angioplasty (PTA) and stenting
* Patients must be at least 18 years of age
* Patient with a life expectance of at least 12 months
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in the following study protocol
* Patients must agree to undergo at least the 6-month clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial, e.g. balloon angioplasty by means of other suitable stent devices. Patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.
* Lesions with unsatisfying angiographic results due to recoil and/or dissections after POBA/DCB interventions
* Infra-inguinal lesions in the superficial femoral artery (SFA) and popliteal segments (P1,P2 & P3) reference vessel diameters between 4 and 7.0 mm, lesion length suitable for the release of at least 2 Stent (up to 6) segments implanted with a minimum inter-stent distance of 1 cm
* Diameter stenosis pre-procedure must be larger or equal to 70%
* Vessels must have adequate distal run-off with at least one vessel to the foot or with collaterals in the calf supplying sufficient flow to the foot.

(Lesions separated by less than 2 cm are considered as one lesion)

Exclusion Criteria:

* Patient not suitable for revascularization by interventional means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of the study is to assess the safety and efficacy of the Multi-LOC® peripheral stent system to treat de novo and restenotic lesions (no in-stent restenosis (ISR), no restenosis post drug coated balloon (DCB)) after flow limiting plain old balloon angioplasty (POBA) and/or DCB dilatations in the superficial femoral artery (SFA) and popliteal segments (P1, P2 & P3)
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
target lesion revascularization | 6 months
  target lesion revascularization surgical & interventional

SECONDARY OUTCOMES:
pain free walking distance | < 3 weeks, 6 months, 12 months
  pain free walking distance
maximum walking distance | < 3 weeks, 6 months, 12 months
  maximum walking distance
target lesion revascularization | 12 months
  target lesion revascularization
procedural success | immediately after Multi-LOC implantation (within the first 30 minutes)
  procedural success to pass and treat the target lesion
ankle brachial index | < 3 weeks, 6 months, 12 months
  ankle brachial index
patency rates | 6 and 12 months
  patency rates observed using non-invasive Duplex ultrasound
Rutherford classification | baseline, < 3 weeks, 6 months, 12 months
  Rutherford classification
Rutherford classification shift | < 3 weeks, 6 months, 12 months
  difference in Rutherford classification compared to previous time point
amputation rate | 6 and 12 months
  rate of major and minor amputations
quality of life assessment | 6 and 12 months
  quality of life assessment through validates CRF's

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Amendt, MD, Principal Investigator — Deaconess Hospital Mannheim
Locations (1):
- Diakonissenkrankenhaus Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sigl M, Beschorner U, Zeller T, Waliszewski M, Langhoff R, Tautenhahn J, Amendt K. Focal Stenting of Complex Femoropopliteal Lesions with the Multi-LOC Multiple Stent Delivery System: 12-Month Results of the Multicenter LOCOMOTIVE Study. Cardiovasc Intervent Radiol. 2019 Feb;42(2):169-175. doi: 10.1007/s00270-018-2095-9. Epub 2018 Oct 25. PMID 30361959